CLINICAL TRIAL: NCT00313599
Title: A Phase I Dose Escalation Study of a 2 Day Oral Lapatinib Chemosensitization Pulse Given Prior To Weekly Intravenous Abraxane™ in Patients With Advanced Solid Tumors
Brief Title: Lapatinib and Paclitaxel in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF CC#05591
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Bladder Cancer; Brain and Central Nervous System Tumors; Breast Cancer; Esophageal Cancer; Extragonadal Germ Cell Tumor; Gastric Cancer; Lung Cancer; Ovarian Cancer; Prostate Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent prostate cancer; stage IV prostate cancer; recurrent bladder cancer; stage IV bladder cancer; recurrent gastric cancer; stage IV gastric cancer; recurrent esophageal cancer; stage IV esophageal cancer; recurrent ovarian germ cell tumor; stage IV ovarian germ cell tumor; adult central nervous system germ cell tumor; ovarian choriocarcinoma; ovarian dysgerminoma; ovarian embryonal carcinoma; ovarian yolk sac tumor; ovarian mixed germ cell tumor; recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent extragonadal non-seminomatous germ cell tumor; recurrent extragonadal seminoma; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; recurrent extragonadal germ cell tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms; Central Nervous System Neoplasms; Breast Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Dysgerminoma; Carcinoma, Ovarian Epithelial | interventions — Lapatinib; Paclitaxel; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib and Paclitaxel (Experimental): Lapatinib will be self-administered orally on days 1 and 2 of weeks 1, 2, and 3 of a 4-week cycle. Lapatinib is the experimental therapy and is being administered using a dose escalation design guided by careful monitoring of toxicities. Abraxane will be administered IV weekly on day 3 of weeks 1, 2, and 3 of a 4-week cycle. Abraxane is being administered at the well tolerated and effective standard dose and schedule of 100mg/m2 weekly 3 out of 4 weeks as defined by previous phase I and II studies. Patients will continue on therapy as long as they are not experiencing toxicities and there is no evidence of disease progression.
  Interventions: Drug: lapatinib; Drug: paclitaxel

INTERVENTIONS:
Drug: lapatinib
  Other Names: Tykerb; Tyverb; lapatinib ditosylate
Drug: paclitaxel
  Other Names: paclitaxel albumin-stabilized nanoparticle formulation; Abraxane; Taxol

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Lapatinib may help paclitaxel work better by making tumor cells more sensitive to the drug. Lapatinib may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving lapatinib together with paclitaxel may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lapatinib when given together with paclitaxel in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of a 2-day pulse of lapatinib that can be given prior to paclitaxel (albumin-stabilized nanoparticle formulation ) (ABI-007; Abraxane™) in patients with advanced solid tumor malignancies.

Secondary

* Define the toxicity of this regimen.
* Determine, preliminarily, the antitumor efficacy and safety of ABI-007 when preceded by a 2-day pulse of lapatinib.
* Characterize the potential of the molecular markers within circulating tumor cells as markers of response (e.g., HER2 and AKT) or apoptotic markers.
* Determine whether lapatinib given at MTD prior to ABI-007 alters the pharmacokinetic properties of the paclitaxel component of ABI-007.

OUTLINE: This is a does-escalation study of lapatinib. Patients are stratified according to dose level.

Patients receive oral lapatinib on days 1, 2, 8, 9, 15, and 16 and paclitaxel (albumin-stabilized nanoparticle formulation) (ABI-007; Abraxane™) IV over 30 minutes on days 3, 10, and 17. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of lapatinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicities.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor, including the following tumor types:

  * Breast cancer
  * Non-small cell lung cancer
  * Prostate cancer
  * Bladder cancer
  * Gastroesophageal junction cancer
  * Ovarian cancer
  * Germ cell tumor
* Advanced or metastatic disease
* No effective curative therapy exists
* Evaluable disease

  * Measurable disease not required
  * Bone-only disease allowed
* No progressing brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious intercurrent medical or psychiatric illness
* No serious active infection
* No gastrointestinal tract disease that would impair a patient's ability to take oral medication
* No history of significant cardiac disease, including any of the following:

  * Congestive heart failure
  * Symptomatic cardiac arrhythmias
  * Unstable angina
* No pre-existing peripheral neuropathy ≥ 2

PRIOR CONCURRENT THERAPY:

* Any number of prior therapies allowed
* Prior paclitaxel, tyrosine kinase inhibitor therapy, or endothelial growth factor inhibitors allowed
* At least 14 days since prior and no concurrent CYP3A4 inducers or herbal or dietary supplements
* At least 7 days since prior and no concurrent CYP3A4 inhibitors
* At least 6 months since prior and no concurrent amiodarone
* More than 1 month since prior chemotherapy, radiotherapy, hormonal therapy, or investigational anticancer agents
* Concurrent continued use of gonadal suppression agents (i.e., goserelin acetate or leuprolide acetate) allowed
* No antacids 1 hour before and after study drug administration
* No concurrent retinoids
* No concurrent hormonal anticancer agent
* No other concurrent anticancer chemotherapy or investigational anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of lapatinib in course 1 | estimated to be 12 weeks

SECONDARY OUTCOMES:
Toxicity | up to 12 weeks
Anti-tumor efficacy and safety every 8 weeks | until disease progression estimated to be 12 weeks
Pharmacokinetics during the first 2 weeks of treatment | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark M. Moasser, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Result] Chien AJ, Illi JA, Ko AH, Korn WM, Fong L, Chen LM, Kashani-Sabet M, Ryan CJ, Rosenberg JE, Dubey S, Small EJ, Jahan TM, Hylton NM, Yeh BM, Huang Y, Koch KM, Moasser MM. A phase I study of a 2-day lapatinib chemosensitization pulse preceding nanoparticle albumin-bound Paclitaxel for advanced solid malignancies. Clin Cancer Res. 2009 Sep 1;15(17):5569-75. doi: 10.1158/1078-0432.CCR-09-0522. Epub 2009 Aug 25. PMID 19706807